CLINICAL TRIAL: NCT04739514
Title: Development of Dysphagia Protocol in Ankara City Hospital Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nazife Kapan (Other)
Responsible Party: Sponsor-Investigator, Nazife Kapan, principal investigator, Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AŞH-NK-TEZ
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild dysphagia (Active Comparator)
  Interventions: Other: Exercises for dysphagia rehabilitation
- Moderate dysphagia (Active Comparator)
  Interventions: Other: Exercises for dysphagia rehabilitation
- Severe dysphagia (Active Comparator)
  Interventions: Other: Exercises for dysphagia rehabilitation

INTERVENTIONS:
Other: Exercises for dysphagia rehabilitation — Diet modifications, postural exercises, compensatory exercises, swallowing exercises

SUMMARY:
Stroke, also called cerebrovascular disease, is a sudden-onset neurological disorder that causes a regional or general dysfunction in the brain due to vascular causes. Dysphagia, one of the common complications of stroke, is associated with increased morbidity and mortality.The aim of this study is to evaluate the clinical evaluation of swallowing in stroke patients and to determine the factors affecting the severity and prognosis of dysphagia in patients with dysphagia.Fifty-five patients with acute stroke and dysphagia who were admitted to Ankara City Hospital Neurology Clinic and diagnosed with stroke by neurology and who did not meet the exclusion criteria will be included in this study. When the patients are admitted to the neurology clinic and will be discharged, they will be evaluated three times, in the first month after discharge.

DETAILED DESCRIPTION:
Stroke, also called cerebrovascular disease, is a sudden-onset neurological disorder that causes a regional or general dysfunction in the brain due to vascular causes. Dysphagia, one of the common complications of stroke, is associated with increased morbidity and mortality.The aim of this study is to evaluate the clinical evaluation of swallowing in stroke patients and to determine the factors affecting the severity and prognosis of dysphagia in patients with dysphagia.Fifty-five patients with acute stroke and dysphagia who were admitted to Ankara City Hospital Neurology Clinic and diagnosed with stroke by neurology and who did not meet the exclusion criteria will be included in this study. When the patients are admitted to the neurology clinic and will be discharged, they will be evaluated three times, in the first month after discharge. Clinical evaluations will be made by the responsible investigator in the examination room. Patients will be evaluated with a bedside swallowing screening test. Patients will be divided into 3 groups as mild, moderate and severe dysphagia according to the test. The patients will be evaluated while they are in the neurology clinic and 1 month after the treatment is given.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute stroke by neurology
* Having trouble swallowing
* 18-85 years old, volunteers

Exclusion Criteria:

* Unconscious
* Uncooperative
* Those with oropharyngeal structural damage
* Patients with malignancies involving the head and neck region

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Gugging swallowing screening test | Change from Baseline Gugging swallowing screening test at 1 months
  The gugging test is a validated test in the assessment of bedside swallowing. This test was defined as 20 points (no dysphagia), 15-19 (mild dysphagia), 10-14 (moderate dysphagia) and 9 points or less (severe dysphagia).
Eating assessment tool-10 | Change from Baseline Gugging swallowing screening test at 1 months
  The eating assessment tool-10 is a test that evaluates dysphagia symptoms and severity without any food intake. This test is a test consisting of 10 questions in total and scoring the questions between "no problem" and "serious problem". As the score increases, the severity of dysphagia increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Şehir Hastanesi, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Broadley S, Cheek A, Salonikis S, Whitham E, Chong V, Cardone D, Alexander B, Taylor J, Thompson P. Predicting prolonged dysphagia in acute stroke: the Royal Adelaide Prognostic Index for Dysphagic Stroke (RAPIDS). Dysphagia. 2005 Fall;20(4):303-10. doi: 10.1007/s00455-005-0032-y. PMID 16633876
- [Result] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885